CLINICAL TRIAL: NCT03343145
Title: A Randomized, Open-label, Active-controlled, Multi-center, Phase III Study to Evaluate the Efficacy, Safety and Immunogenicity of Leucostim® Versus Neupogen® in Breast Cancer Patients Receiving Myelosuppressive Chemotherapy
Brief Title: A Study to Evaluate the Efficacy, Safety and Immunogenicity of Leucostim® Versus Neupogen® in Breast Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DAGCSF_NP_III
Record Dates: First submitted 2017-11-10; First posted 2017-11-17 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Breast Cancer
Keywords: Neutropenia
MeSH Terms: conditions — Breast Neoplasms; Neutropenia | interventions — Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Drug Group (Experimental): Leucostim 5µg/kg/day
  Interventions: Biological: Leucostim 5µg/kg/day
- Reference Drug Group (Active Comparator): Neupogen 5µg/kg/day
  Interventions: Biological: Neupogen 5µg/kg/day

INTERVENTIONS:
Biological: Leucostim 5µg/kg/day — 5µg/kg/day (based on actual body weight) Leucostim®, subcutaneously, once a day, for up to 14 days or until the target ANC of 10,000/mm3 following the expected chemotherapy-induced ANC nadir
  Arms: Test Drug Group
Biological: Neupogen 5µg/kg/day — 5µg/kg/day (based on actual body weight) Neupogen®, subcutaneously, once a day, for up to 14 days or until the target ANC of 10,000/mm3 following the expected chemotherapy-induced ANC nadir
  Arms: Reference Drug Group

SUMMARY:
A study to compare the efficacy, safety and immunogenicity of Leucostim® to those of Neupogen® in patients with breast cancer intended to be treated with TAC regimen as a myelosuppressive chemotherapy.

DETAILED DESCRIPTION:
TAC regimen (docetaxel, doxorubicin and cyclophosphamide) is recommended for the adjuvant treatment of breast cancer patients. The TAC regimen is known to lead to significant hematological toxicity and induces febrile neutropenia with a rate > 20%. The use of primary G-CSF prophylaxis with the TAC regimen is recommended by guidelines. e.g., by the European Organisation for Research and Treatment of Cancer as well as by the guideline on myeloid growth factors of the National Comprehensive Cancer Network.6,7 This study is to compare the efficacy, safety and immunogenicity of Leucostim® to those of Neupogen® in patients with breast cancer intended to be treated with TAC regimen as a myelosuppressive chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to provide a written informed consent
2. Men or women ≥ 18 and ≤ 70 years of age
3. Histologically or cytologically confirmed breast cancer (Stage II to Stage IV)
4. Be scheduled to receive TAC regimen as adjuvant therapy
5. Subjects who meet the conditions at screening test as follows;

   * Absolute Neutrophil Count (ANC) ≥ 1,500/mm3
   * Platelet Count ≥ 100,000/mm3
   * ECOG Performance Status : 0~2
6. Adequate renal function (Creatinine ≤ 1.5 x ULN at screening test)
7. Adequate hepatic function at screening test (Total bilirubin/AST/ALT ≤ 1.5 x ULN, ALP ≤ 2.5 x ULN at screening test)

Exclusion Criteria:

1. Prior chemotherapy experiences
2. Prior bone marrow or stem cell transplantation
3. History of treatment with hematopoietic growth factors (e.g. G-CSF, peg-G-CSF, erythropoietin)
4. History of prior malignancy other than breast cancer or surgically cured malignancies within 5 years of informed consent date
5. Participation in any other clinical study within 4 weeks of informed consent date or planning to simultaneously participate in another clinical study
6. Currently receiving radiation therapy or having completed radiation therapy within 4 weeks of informed consent date
7. Active infection which may require systemic antimicrobial or antiviral therapy during the study (e.g. ANC ≥ 12,000/mm3 or Body Temperature > 38.2 degrees C (100.8 degrees F))
8. History of systemic antibiotic use within 72 hours prior to chemotherapy
9. History of hypersensitivity to the investigational product, components or similar products
10. HIV positive
11. Pregnant or lactating women, or women of child-bearing potential who are not willing to follow a reliable and effective contraceptive measure during the course of the study and for at least one month after the completion of the study
12. Any other cases that is considered by the investigator as an exclusion

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2017-01-12 (Actual); Primary Completion 2019-01-28 (Actual); Study Completion 2019-07-29 (Actual)

PRIMARY OUTCOMES:
Mean duration of Grade 4 Neutropenia (i.e. ANC < 500/mm3) in Cycle 1 | Maximum of 14 Days

SECONDARY OUTCOMES:
Depth of ANC nadir after chemotherapy in Cycle 1 | Maximum of 14 Days
Time to ANC recovery in Cycle 1 | Maximum of 14 Days
Incidence of febrile neutropenia in Cycle 1; | Maximum of 14 Days

OTHER OUTCOMES:
Anti-rhG-CSF antibody formation | 180±14d

CONTACTS AND LOCATIONS:
Locations (1):
- RSUP Dr. Hasan Sadikin, Bandung, Indonesia

IPD SHARING:
Plan to Share IPD: No